CLINICAL TRIAL: NCT01178385
Title: Cognitive-Behavioral Treatment for Anxiety Disorders in Children With Autism Spectrum Disorders
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACH-2010
Record Dates: First submitted 2010-08-05; First posted 2010-08-10 (Estimated); Results first posted 2013-04-02 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2012-12

CONDITIONS: Autism; Asperger's Syndrome; Generalized Anxiety Disorder; Social Phobia; Separation Anxiety Disorder; Obsessive-compulsive Disorder
Keywords: Autism; Asperger's Syndrome; Treatment; Cognitive-behavioral therapy; Anxiety; Children; Therapy
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome; Generalized Anxiety Disorder; Phobia, Social; Anxiety, Separation; Obsessive-Compulsive Disorder; Anxiety Disorders | interventions — Cognitive Behavioral Therapy; Psychotherapy; Counseling; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-behavioral therapy (Experimental): Therapists will work with families for 16 weekly sessions implementing the Behavioral Interventions for Anxiety in Children with Autism (BIACA) CBT program, which is a modified version of a family CBT treatment manual for typically developing children with anxiety disorders. The BIACA intervention program is flexible in nature and employs a modular format. Despite the added flexibility of the modular format, a minimum of three sessions are spent on basic coping skills and eight are spent on in vivo exposure to ensure an adequate and comparable dose of the core elements of CBT for anxiety across cases.
  Interventions: Behavioral: Cognitive-behavioral therapy
- Treatment as Usual (Active Comparator): Participants randomized to this arm will be instructed to continue receiving their prior interventions as recommended by their providers (e.g., psychotherapy, social skills training, behavioral interventions, family participation in family therapy or a parenting class, or pharmacological interventions). Treatment changes (e.g., medication increase, starting psychotherapy in the community) are not prohibited and will be monitored. Thus, treatment will continue as it would in standard practice; and will be monitored through periodic study assessment.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — Therapists will work with families for 16 weekly sessions implementing the Behavioral Interventions for Anxiety in Children with Autism (BIACA) CBT program, which is a modified version of a family CBT treatment manual for typically developing children with anxiety disorders. The BIACA intervention program is flexible in nature and employs a modular format. Despite the added flexibility of the modular format, a minimum of three sessions are spent on basic coping skills and eight are spent on in vivo exposure to ensure an adequate and comparable dose of the core elements of CBT for anxiety across cases.
  Other Names: psychotherapy; counseling; therapy
  Arms: Cognitive-behavioral therapy
Behavioral: Treatment as Usual — Participants randomized to this arm will be instructed to continue receiving their prior interventions as recommended by their providers (e.g., psychotherapy, social skills training, behavioral interventions, family participation in family therapy or a parenting class, or pharmacological interventions). Treatment changes (e.g., medication increase, starting psychotherapy in the community) are not prohibited and will be monitored. Thus, treatment will continue as it would in standard practice; and will be monitored through periodic study assessment.
  Arms: Treatment as Usual

SUMMARY:
Autism spectrum disorders affect as many as 1 out of 150 children and are related to significant impairment in social, adaptive, and school functioning. Co-occurring conditions, such as anxiety, are common and may cause substantial distress and impairment beyond that caused by the autism diagnosis. Although effective interventions have been developed for typically developing youth with anxiety disorders, this approach needs to be adapted for children with autism. Accordingly, we are proposing a randomized controlled trial to examine the effectiveness of CBT relative to treatment as usual (TAU) in 46 youth ages 7-11 with autism spectrum disorders and comorbid anxiety disorder(s).

DETAILED DESCRIPTION:
Autism spectrum disorders affect as many as 1 out of 150 children (Centers for Disease Control, 2007), with many higher-functioning children not being diagnosed until elementary school or later (Fombonne, 2003). Significant impairment in social, adaptive, and school functioning is prevalent and longstanding (Howlin et al., 2004). In addition, comorbid psychological disorders are common in the ASD population (Simonoff et al., 2008), and may cause substantial distress and impairment beyond that caused by the ASD diagnosis. Comorbid anxiety disorders, in particular, affect as many as 80% of children and adolescents with ASD (Bellini, 2004; de Bruin et al., 2007; Klin et al., 2005; Muris et al., 1998). Although efficacious interventions have been developed for otherwise typically developing youth with anxiety disorders, the linguistic; cognitive; and social characteristics of ASD may render standard treatment approaches less effective for children with ASD (Volkmar & Klin, 2000). Thus, there is a clinical need for the modification of existing treatment modalities for this unique group. To date, few studies have experimentally tested the efficacy of CBT for youth with a comorbid presentation of anxiety and ASD. This gap in the literature is of particular concern given the prevalence of comorbid anxiety among children, consequences of untreated anxiety, unknown efficacy of antidepressant medication for anxiety in ASD, and potential safety and tolerability issues related to medication use. Accordingly, we are proposing a randomized controlled trial to examine the efficacy of CBT relative to treatment as usual (TAU) in 46 youth ages 7-11 with ASD and comorbid anxiety disorder(s). In the proposed grant, we will: (1) examine the acute efficacy of CBT relative to TAU, and (2) evaluate the short-term maintenance of treatment gains. Forty-six children (ages 7-11 years) with ASD and comorbid anxiety disorder(s) will be randomly assigned to one of the two treatment conditions. Primary outcomes will be assessed by an independent evaluator, and will include change in anxiety symptom severity; response rates; and remission rates. Considering the rising number of children diagnosed with ASD, our proposed work toward the advent of an efficacious CBT protocol will provide a timely contribution to public health efforts.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient children with an autism spectrum disorder (see #2 below) between the ages 7-11years.
2. Meets criteria for a diagnosis of autism, Asperger syndrome (AS), or PDD-NOS using scores from the Autism Diagnostic Interview-Revised and Autism Diagnostic Observation Schedule.
3. Meets DSM-IV criteria for a diagnosis of one of the following anxiety disorders: separation anxiety disorder (SAD), generalized anxiety disorder (GAD), social phobia, or obsessive compulsive disorder (OCD) as determined by the ADIS-IV-C/P (with CSR 4) and all available information.
4. Minimum score of 14 on the PARS Severity Scale; this score indicates clinically significant anxiety symptom severity (RUPP, 2002) and has been used in recent major clinical trials (e.g., Walkup et al., 2008).
5. Child has a Full Scale and Verbal Comprehension IQ > 70 as assessed on a commonly used IQ test.
6. Subjects with co-morbid depression, ADHD, tic disorder or disruptive behavior disorders will be acceptable as long as the anxiety disorder is primary (i.e., most impairing/distressing).

Exclusion Criteria:

1. Receiving concurrent psychotherapy, social skills training, or behavioral interventions (e.g., applied behavior analysis). Families will have the option of discontinuing such services to enroll in the study. Those randomized to TAU will be able to continue or initiate psychosocial interventions (psychotherapy, social skills training, applied behavior analysis, or family therapy) whereas those randomized to CBT will not receive these interventions concurrent with CBT.
2. New Treatments: Initiation of an antidepressant within 12 weeks before study enrollment or an antipsychotic 8 weeks before study enrollment. No new alternative medications, nutritionals or therapeutic diets within 8 weeks of study enrollment.
3. Established Treatment changes: Any change in established psychotropic medication (e.g., antidepressants, anxioloytics) within 8 weeks before study enrollment, or any change in alternative medications that might have behavioral effects within 6 weeks prior to the study baseline assessment. Those randomized to TAU may make medication changes following randomization, including starting a medication; those randomized to CBT will remain stable on medications during the study.
4. (a) Current clinically significant suicidality or (b) individuals who have engaged in suicidal behaviors within 6 months will be excluded and referred for appropriate clinical intervention.
5. Lifetime DSM-IV bipolar, schizophrenia or schizoaffective disorders; or Substance abuse in past 6 months.
6. Unwillingness of parents to make the commitment to accompany their child for multiple study visits.
7. Presence of a significant and/or unstable medical illness which might lead to hospitalization during the study.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Storch, Ph.D., Principal Investigator — University of South Florida
Locations (1):
- Rothman Center for Neuropsychiatry, University of South Florida, St. Petersburg, Florida, United States

REFERENCES:
- [Derived] Storch EA, Arnold EB, Lewin AB, Nadeau JM, Jones AM, De Nadai AS, Jane Mutch P, Selles RR, Ung D, Murphy TK. The effect of cognitive-behavioral therapy versus treatment as usual for anxiety in children with autism spectrum disorders: a randomized, controlled trial. J Am Acad Child Adolesc Psychiatry. 2013 Feb;52(2):132-142.e2. doi: 10.1016/j.jaac.2012.11.007. Epub 2013 Jan 2. PMID 23357440

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-five children between 7-11 years (M=8.89, SD=1.34) were recruited through referrals, advertisements, and the patient flow at a university-based mental health clinic. Recruitment took place between March, 2010 and ended around January, 2012.
Pre-assignment Details: Seventy-one youth were assessed for eligibility. Twenty-six were excluded because they did not meet eligibility criteria (Did not meet IQ criteria (n=6); Did not meet anxiety criteria (n=9); Parent unwilling or unable to accompany child to all sessions (n=4); No autism spectrum disorder diagnosis (n=7)).
Period: Overall Study
Arm/Group | Cognitive-behavioral Therapy | Treatment as Usual
Started | 24 | 21
Completed | 22 | 21
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive-behavioral Therapy | Treatment as Usual | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 21 | 45
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 8.83 (1.31) | 8.95 (1.40) | 8.89 (1.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 19 | 17 | 36
Region of Enrollment [Number; unit: participants]
  United States | 24 | 21 | 45

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Anxiety Rating Scale (Measures the Severity of Anxiety Symptoms)
Description: This scale assesses the severity of anxiety symptoms. The scale ranges from 0 (minimum score) to 25 (maximum score). Higher scores reflect more severe anxiety symptoms; lower scores reflect lower anxiety severity. There are no subscales to this measure.
Time Frame: After an average of 16 weeks (Post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy | Treatment as Usual
Number analyzed (Participants) | 24 | 21
units on a scale
  Baseline | 16.33 (1.93) | 17.62 (2.04)
  Post-treatment | 11.58 (3.15) | 16.05 (3.22)

2. Secondary Outcome: Anxiety Disorders Interview Schedule Highest Anxiety Clincian Severity Rating (Measures the Severity of the Child's Anxiety Symptoms)
Description: This is a measure of severity of the child's primary anxiety disorder. The maximum rating is 8, the minimum rating is 0. Higher scores correspond to more severe anxiety.
Time Frame: After an average of 16 weeks (Post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy | Treatment as Usual
Number analyzed (Participants) | 24 | 21
units on a scale
  Baseline | 5.42 (.72) | 5.62 (.92)
  Post-treatment | 3.38 (1.81) | 4.9 (1.51)

3. Secondary Outcome: Clinical Global Impression - Severity Scale (This Scale Measures the Severity of the Child's Anxiety Symptoms).
Description: This scale measures severity of the child's overall anxiety presentation. The minimum rating is 0, the maximum is 6. Higher scores correspond to greater anxiety; lower scores correspond to less severe anxiety. There are no subscales for this measure.
Time Frame: After an average of 16 weeks (Post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy | Treatment as Usual
Number analyzed (Participants) | 24 | 21
units on a scale
  Baseline | 3.5 (.72) | 4 (.63)
  Post-treatment | 2.67 (.48) | 3.57 (.87)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: During the course of the acute intervention (16 weeks duration).
Arm/Group | Cognitive-behavioral Therapy | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
1. Modest sample size was modest.
2. Only ~75% of families in the treatment as usual arm had some form of active intervention.
3. Short follow-up interval that only included treatment responders in the CBT arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No